CLINICAL TRIAL: NCT06979245
Title: Validity and Reliability in Turkish of Vascular Quality of Life Questionnaire-6 in Patients Diagnosed With Takayasu Arteritis and Vascular Behçet's Disease
Brief Title: Turkish Adaptation of the VascuQoL-6 Quality of Life Scale
Status: Completed | Type: Observational
Sponsor: Uşak University (Other)
Collaborators: Pamukkale University (Other)
Responsible Party: Principal Investigator, Kevser Gürsan, Principal Investigator, Uşak University
Other Study IDs: E-60116787-020-494225
Record Dates: First submitted 2025-05-11; First posted 2025-05-18 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Takayasu Arteritis; Behcet Disease; Quality of Life
Keywords: Takayasu arteritis; Behcet Disease; Turkish; Validity; Reliability; Quality of life
MeSH Terms: conditions — Takayasu Arteritis; Behcet Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Those diagnosed with Takayasu Arteritis or Vascular Behçet's disease: The study group was diagnosed with Takayasu Arteritis or Vascular Behçet's disease by a rheumatologist.

SUMMARY:
Study type: Observational study Primary objective: The aim of this study was to examine the validity and reliability of the Vascular Quality of Life Questionnaire-6 (VascuQoL-6) in Turkish in individuals diagnosed with Takayasu Arteritis or Vascular Behçet's disease.

The main questions it aims to answer are:

Can VascuQoL-6 measure disease-related quality of life validly and reliably? Does the scale show significant correlations with measures such as SF-36, EQ-5D-3L, BDCAF, BSAS and ITAS-2010? There is no comparison group.

Participants will be asked to:

Contribute to the translation process of the scale into Turkish, Complete all quality of life forms in the first assessment, Participate in the test-retest analysis by re-filling VascuQoL-6 one week later.

DETAILED DESCRIPTION:
Takayasu arteritis (TA) is a rare, systemic granulomatous large vessel vasculitis that primarily affects the aorta and its branches. Although all major arteries can be affected, the descending and ascending aorta, subclavian arteries, and carotid arteries are most commonly affected. Inflammation can lead to intimal proliferation and stenosis or destruction of the vascular structure and aneurysmal degeneration. TA is a disease with profound consequences on quality of life.

Behçet's disease is a multisystemic, chronic inflammatory vasculitis characterized by skin and mucosal lesions.

The vascular involvement of Behçet's disease has characteristic features. The most important difference between Behçet's disease and other vasculitides is that venous involvement is more prevalent than arterial involvement. Many different symptoms can coexist with vascular involvement, and these symptoms require different treatments. BD characterized by vascular involvement may be a cluster different from the typical clinical setting and may differ from the typical symptomatic group in terms of treatment resistance and prognosis.

It is recommended that objective outcome measures be complemented by patient-reported outcome measures. Such measures, when integrated into daily clinical practice, are useful in clinical decision making and can also provide important information about the results of different interventions. Therefore, it is widely recommended to use disease-specific health-related quality of life instruments. Because outcome measures that focus on the specific limitations experienced by patients are made sensitive to detecting significant changes in health status in response to treatment. The Vascular Quality of Life (VascuQoL) questionnaire was developed by Morgan et al in 2001 and has been translated into 7 languages.

The aim of this study was to examine the validity and reliability of the Turkish version of the Vascular Quality of Life Questionnaire-6 in patients diagnosed with Takayasu Arteritis and Vascular Behçet's disease.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-65
* Being willing to participate in the study
* Being diagnosed with Takayasu Arteritis or Vascular Behçet's disease by a rheumatologist

Exclusion Criteria:

* Having another disease that will affect their physical condition
* Having a cognitive disability that will prevent them from cooperating
* Being pregnant
* Having a neurological disease (hemiplegia, Parkinson's, multiple sclerosis, vertigo, epilepsy, etc.)
* Having undergone any surgery in the last year
* Having another simultaneous rheumatic disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Those diagnosed with Takayasu Arteritis or Vascular Behçet's disease
Sampling Method: Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-08-10 (Actual); Study Completion 2025-08-10 (Actual)

PRIMARY OUTCOMES:
Vascular Quality of Life Questionnaire-6 | At enrollment and 1 week
  VascuQoL aims to assess quality of life in peripheral arterial disease, regardless of disease severity (i.e. in intermittent claudication and critical limb ischemia). It consists of 6 items. Each item has a 7-point response scale (1: worst quality of life; 7: best quality of life).

SECONDARY OUTCOMES:
Takayasu Arteritis: Kerr Criteria and Indian Takayasu's Clinical Activity Score (ITAS2010) | At enrollment
  In Takayasu arteritis, the disease extent index (DEI.TAK) was developed in TAK as a criterion that focuses on findings related to large vessel disease rather than general characteristics of the disease. In 2010, the new version of DEI.TAK, the Indian Takayasu Clinical Activity Score-ITAS2010, was created. The 5 main items belonging to the cardiovascular (CV) system, Hypertension and Stroke, are scored as 2 points each. All other items (marked only as circles) are scored as 1 point each. In addition to the 2 points due to the presence of the first 5 items in the CV section, each murmur, claudication, loss of pulse or pulse inequality is scored as 1 point each, and the total score is determined by adding these 2 points. When calculating the acute phase response ITAS (ITAS.A), first the ITAS2010 is calculated and then the acute phase response values are scored as 1-3 points within certain intervals and added to the ITAS2010 score. The definition of active disease is > 1 point for ITAS2
Short Form-36 | At enrollment
  It is one of the most frequently used scales to measure quality of life, consisting of 8 subcategories: physical functionality, social functionality, role limitations due to physical complaints, role limitations due to emotional problems, mental health, energy-vitality, pain, and general health perception. Separate scores are obtained for each subscale and the scores range from 0 to 100. A score of 100 indicates good health status, and a score of 0 indicates poor health status. Its Turkish validity was carried out by Koçyiğit et al. in 1999.
EQ-5D-3L General Quality of Life Scale | At enrollment
  EQ-5D-3L consists of two parts: EQ-5D-3L descriptive system and EQ-5D-3L visual analog scale (EQ-5D-3L VAS). EQ-5D-3L descriptive system total score is between -0.59 and 1. "1" indicates the best health, while negative values indicate low quality of life. EQ-5D-3L VAS is scored between "0" and "100". (0: worst imaginable health status and 100: best imaginable health status)
Behcet's Disease Current Activity Form (BDCAF) | At enrollment
  This index aims to evaluate all types of involvement in Behçet's disease. BDCAF is filled out by the clinician and the evaluation is made considering the day the patient comes and the last 4 weeks. The evaluation of major organ involvements such as eye, gastrointestinal system and neurological involvement should be done by experts in their field. Active findings seen in the last 4 weeks in all systems are scored and a score between 0 and 12 is obtained.It has been stated that the BDCAF score must be 2 or above for the disease to be considered active.
Behçet Syndrome Activity Scale | At the enrollment
  Unlike BDCAF, it is completely filled out by the patient. Similar to BDCAF, the last 4 weeks are evaluated. It is a form consisting of a total of 10 questions that can be filled out very quickly. The first 6 questions are about mucocutaneous involvement, and the other questions ask about eye, gastrointestinal and vascular involvement. Its advantage is that it also asks how much each lesion bothers the patient. However, there is no weighting according to the types of involvement in this index as in BDCAF.

CONTACTS AND LOCATIONS:
Overall Officials: Bilge Basakcı Calık, Prof. Dr., Principal Investigator — Pamukkale University
Locations (2):
- Turkey (Türkiye) (2):
  - Pamukkale University Rheumatology Clinic and Pamukkale University Faculty of Physiotherapy and Rehabilitation, Denizli
  - Pamukkale University, Denizli

IPD SHARING:
Plan to Share IPD: No
In order to protect participant confidentiality and comply with the confidentiality commitment approved by the ethics committee, no sharing of individual-level data is planned. In addition, the ethics committee decision that approved the study covers data use with limited access only. Therefore, it may not be possible to share IPD data publicly.